CLINICAL TRIAL: NCT06227221
Title: A Phase 2, Randomized, Placebo Controlled Study Investigating the Efficacy and Safety of Sorafenib in New-Onset Type 1 Diabetes Mellitus
Brief Title: Efficacy and Safety of Sorafenib in New-Onset Type 1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023ZLNL001
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Experimental): Subjects receive sorafenib 400mg once daily. Insulin therapy will be continued as a routine therapy.
  Interventions: Drug: Sorafenib
- Placebo (Placebo Comparator): Subjects receive placebo 400mg once daily. Insulin therapy will be continued as a routine therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib — Subjects receive sorafenib 400mg once daily. Insulin therapy will be continued as a routine therapy.
  Arms: Sorafenib
Drug: Placebo — Subjects receive placebo 400mg once daily. Insulin therapy will be continued as a routine therapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the therapeutic effect and safety of Sorafenib in T1DM patients.

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is caused by autoimmune destruction of beta cells in the islet. Insulin has been used as a routine therapy for T1DM to alleviate the hyperglycemic status, yet cannot effectively prevent the progressing destruction of beta cells or preserve its function. Our preliminary data identified sorafenib as an inhibitor of Th1 differentiation and an indirect inhibitor of JAK2 and found that sorafenib prevented and reversed T1DM in NOD mice by decreasing the accumulation of Th1 cells and the expression of inflammatory cytokines in pancreas. Sorafenib is already in clinical use for renal cell carcinoma, hepatocellular carcinoma and differentiated thyroid cancer. It is hypothesized that sorafenib treatment for 26 weeks will preserve beta cell function in adults with new-onset T1DM. The aim of this study is to investigate the potential of sorafenib on preserving beta cell functions in human T1DM.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with written informed consent;
2. Age: 18-60 years;
3. Diagnosis of T1DM according to ADA criteria within 1 year prior to starting study drug;
4. Islet autoantibody positivity (one or more of GADA, IA-2A, ZnT8A);
5. Stimulated C-peptide > 200 pmol/L;
6. Participants of childbearing age who are sexually active must agree to use of effective birth control until the end of the study

Exclusion Criteria:

1. Non-Type 1 Diabetes Mellitus.
2. Signs of chronic active infection (e.g., hepatitis, tuberculosis, cytomegalovirus, Epstein-Barr virus, herpes zoster, or toxoplasmosis), or screening laboratory evidence consistent with chronic active infection:

   * Positivity for human immunodeficiency virus
   * Positive purified protein derivative or interferon-γ release assay suggestive of tuberculosis
   * Positivity for hepatitis B surface antigen And acute infections (e.g., respiratory, urinary tract, or gastrointestinal infections) must be resolved before reevaluation;
3. Severe hypertension (systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg, or those requiring the concurrent use of 3 or more antihypertensive medications);
4. Previous or current cerebro-cardiovascular diseases:

   * Congestive heart failure (NYHA Class III-IV)
   * Myocardial infarction
   * unstable ischemic heart disease,
   * Arrhythmia
   * Syncope of cardiac or unknown origin
   * Structural defects
   * Signs of QT prolongation on electrocardiogram (450 ms in men, 470 ms in women)
   * Stroke
   * Transient Ischemic Attack
5. Hematological conditions:

   * Anemia (hemoglobin below 120 g/L in men and 110 g/L in women)
   * Leukopenia (<4000 leukocytes per μL)
   * Thrombocytopenia (<100,000 platelets per μL)
   * Neutropenia (<1500 neutrophils per μL)
6. Abnormal coagulation function during the screening period: Prothrombin time (PT) is prolonged beyond the upper limit of normal for 3 seconds and/or activated partial thromboplastin time (APTT) is prolonged beyond the upper limit of normal for 10 seconds;
7. Liver and renal dysfunction:

   * acute or chronic active hepatitis
   * alanine aminotransferase or aspartate aminotransferase >2·0 times the upper limit of normal persisting for persisting for more than one week
   * impaired renal function defined by estimated glomerular filtration rate (according to the CKD-EPI) of < 60 mL/min/1.73 m2
8. History of severe gastrointestinal diseases such as gastrointestinal ulcers, gastrointestinal hemorrhage, pyloric stenosis, gastric bypass surgery, acute or chronic pancreatitis, etc;
9. Have had any major surgery within 8 weeks prior to screening or will require major surgery during the study;
10. Anticipated ongoing use of diabetes medications other than insulin;
11. Known hypersensitivity to sorafenib, or history of severe allergic reactions to other medications (e.g., anaphylaxis, angio-edema, or serious cutaneous drug reactions);
12. Use of medications in the last month known to cause an ongoing change in the course of type 1 diabetes or immunological status (e.g., high-dose inhaled, extensive topical, or systemic glucocorticoids);
13. Previous treatment with sorefenib or related multikinase inhibitor;
14. Concurrent use of medications that affect cytochrome P450 3A4 or use of drugs that interact with sorefenib, leading to altered plasma concentrations of the drugs;
15. For men: unwilling to adopt contraception during the whole study period;
16. For women:

    * Pregnancy or breastfeeding
    * Less than 100 days postpartum before enrollment
    * Unwilling to defer pregnancy during the 1-year study period
17. Known coagulation disorders or use of anticoagulants (e.g., warfarin, rivaroxaban, or low molecular weight heparin);
18. Other situations in which the investigator considers it inappropriate to participate in this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the change from baseline of serum C-peptide area under the curve (AUC) over 2 hours following a mixed meal | Measured at week 26
  The change from baseline of serum C-peptide (pmol/L)

SECONDARY OUTCOMES:
Change from baseline of serum C-peptide area under the curve (AUC) over 2 hours following a mixed meal | Measured at week 52
  Change from baseline of serum C-peptide area under the curve (AUC) over 2 hours following a mixed meal tolerance test
Change from baseline in glycosylated haemoglobin (HbA1c) levels | Measured at weeks 4, 12, 26 and 52
  Change from baseline in HbA1c (%) levels
Change from baseline in insulin dosage | Measured at week 26 and 52
  Change from baseline in insulin dosage, including total dose and units per kilogram
The frequency and severity of hypoglycemic events | Measured at week 26 and 52
  Number and rate of hypoglycemic events including Grade 1, 2 and 3
Drug safety: gastrointestinal symptoms, rashes, fatigue, bleeding, anemia, infections, cardiovascular events, etc. | Measured at week 26 and 52
  Number and rate of gastrointestinal symptoms, rashes, fatigue, bleeding, anemia, infections, cardiovascular events, etc.

IPD SHARING:
Plan to Share IPD: Undecided